CLINICAL TRIAL: NCT04316650
Title: Study of Maintenance of the Efficiency and Adverse Effects of Pharmacological Treatments in Sex Offenders With Paraphilia
Acronym: ESPARA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P150962J; 2017-004984-11 (EudraCT Number)
Record Dates: First submitted 2019-09-02; First posted 2020-03-20 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Paraphilia
Keywords: Paraphilia; SSRI anti-androgen; Psychological treatment; Preservation of efficiency; Pharmacological treatment; Side effects
MeSH Terms: conditions — Paraphilic Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SSRI Group (Other): Treated by ISRS at inclusion
  Interventions: Behavioral: Evaluation Scales; Other: osteodensitometry; Biological: blood samples; Other: ECG; Genetic: Blood and saliva samples
- Anti-androgen Group (Other): Treated by anti-androgen at inclusion
  Interventions: Behavioral: Evaluation Scales; Other: osteodensitometry; Biological: blood samples; Other: ECG; Genetic: Blood and saliva samples
- No SSRIs or antiandrogen treatment at inclusion (Other): no treatment
  Interventions: Behavioral: Evaluation Scales; Other: osteodensitometry; Biological: blood samples; Other: ECG; Genetic: Blood and saliva samples

INTERVENTIONS:
Behavioral: Evaluation Scales — * PATHOS / PEACCE : hypersexuality diagnostic scale
  * PDQ-4+: Personality Diagnostic Questionnaire version 4
  * AUDIT
  * Life trajectory : THQ
  * Cognitive function (MoCA, Stroop)
  * ISDSS: and self report of sexual activity and desire
  * BARS: Brief Adhesion Rating Scale (treatment observance)
  * SF-36 scale : quality of life
  * BDI-II : Beck Depression Inventory
  * BSSI ; Beck suicidal Inventory
  * Cognitive functioning evaluation : Molest and Rape Scale
  * Empathy: EMPAT
  * Evaluation of Cognitive functioning: denial evaluation and Mc Kibben minimization
  * Baratt Impulsivity Scale
  * CSBI
  * Static 99 and Stable 2007
Other: osteodensitometry — Osteodensitometry
Biological: blood samples — * Lipid profile (total cholesterol, triglycerides, HDL cholesterol)
  * Liver function (ASAT, ALAT, total bilirubin, transferase gamma-glutamyl et alcalin phosphatases
  * Kydney function
  * Blood count
  * Biological Measurements and Measurement of Systematic Plasma Testosterone and TeBG Levels in Sex Offenders check for pathology of the Gonadotropin Axis
  * Biological Measurements of Plasma Prolactin level
Other: ECG — ECG (heart rate, search for cardiac conduction disorders or cardiac arrhythmias)
Genetic: Blood and saliva samples — Blood and saliva samples

SUMMARY:
This research concerns the evaluation of the maintenance of the efficiency and incidence of adverse effects of pharmacological treatments in sex offenders with paraphilia.

Despite the increasing use of pharmacological treatments in these indications, there are few data to indicate which sex offender populations benefit from which pharmacological treatments and which adverse events are observed, particularly with anti-androgens or antidepressant treatments that are widely used in these subjects. A recent Cochrane study showed that psychodynamic treatment is less effective in terms of sexual delinquency compared to probation alone and has not shown significant efficacy of cognitive behavioral therapy (CBT) compared to the lack of treatment, except for a study in which anti-androgen therapy was associated with CBT. Another recent study concluded that the tolerance, even of anti-androgenic drugs, was uncertain, as all studies were small and of limited duration, and new research is needed in the future. Further research demonstrating the efficacy of SSRIs in the treatment of paraphilic disorders is still needed and long-term studies are lacking. Their use for this indication is still off label.

As far as we know, this cohort should be the largest population of paraphilic sex offenders studied for the longest time to date in a field where research is insufficient. This large sample receiving routine care and followed for 3 years should allow to analyse the maintenance of the effectiveness of the pharmacological treatments received (SSRIs or anti-androgens), and their tolerance. In addition, this analysis of clinical practices should be crucial to improve the knowledge of the indications for these treatments, which could possibly be reviewed with respect to their effectiveness and tolerance, especially in the most serious cases of paraphilic sex offenders.

DETAILED DESCRIPTION:
This research uses a "naturalistic" follow-up method (over 3 years). The main objectives focuses on two main issues that are important in clinical practice: (1) the tolerance of anti-androgenic treatments traditionally used for many years in young sexual offenders with severe paraphilias (2) the maintenance of the efficiency of SSRIs not yet approved for this indication (despite their current use in the treatment of minor paraphilic disorders).

The paraphilic sex offender population are divided into three groups: those receiving SSRIs, those receiving anti-androgens (either GnRH agonists or CPA) and those receiving no pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

Man

* At least one sex offence
* Paraphilia (DSM-5 criteria )
* Receiving pharmacological treatment ( ISRS or anti-androgen or none of them)
* Age between 18 and 65 years
* Patient 100% covered by social security

Exclusion Criteria:

* no consent
* female
* aged under 18 or over 65 years
* subject receiving simultaneous ISRS and anti-androgen treatment before enrolment
* incarcerated
* Subject under guardianship (patients under curatorship may however be included),
* no social security registration
* contraindications or allergies to treatments

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Sexual desire and activity intensity scale | Change from inclusion at 36 months
  ISRS Group and no pharmacological treatment group : Treatment efficiency : Sexual desire intensity and scale to measure deviant and non deviant sexual behavior symptoms. (Lickert's scale, scale range : 0 to 7)
Incidence of adverse events | 36 months
  Anti-Androgen Group and no pharmacological treatment group : Report of any adverse event: the type, frequency, time of occurrence of adverse events

SECONDARY OUTCOMES:
Sexual desire intensity scale | Every 3 months up to 36 months
  Anti-Androgen Group : Treatment efficiency : Sexual desire intensity and scale to measure deviant and non deviant sexual behavior symptoms
Incidence of adverse events | Every 3 months up to 36 months
  ISRS Group: Report of any adverse event: the type, frequency, time of occurrence of adverse events
Clinical factors | Every 3 months up to 36 months
  All groups : Maintenance of efficacy and incidence of side effects will be analysed taking into account clinical factors listed above.
Psychological factors | Every 3 months up to 36 months
  All groups : Maintenance of efficacy and incidence of side effects will be analysed taking into account psychological factors listed above.
Demographic factors | Every 3 months up to 36 months
  All groups : Maintenance of efficacy and incidence of side effects will be analysed taking into account demographic factors listed above.
Relapse rate | Every 3 months up to 36 months
  Must stay rare event (low expected number, sexual offense risk evaluated in literature around 10%when the treatment is controlled regularly, the relapses are statistically analysed if the numbers is sufficient, but it can not be a principal assessment because of their rarity).

CONTACTS AND LOCATIONS:
Overall Officials: Florence THIBAUT, MD, PhD, Study Chair — CHU Cochin, Groupe Hospitalier Paris Centre
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No